CLINICAL TRIAL: NCT05296551
Title: Examination of a Novel Cognitive-motor Weight-bearing Dual-task Intervention in Older Adults
Brief Title: Dual-task Training in Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruitment within a reasonable timeframe. Primary Investigator has also moved institutions.
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Keith Cole, Assistant Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCR213528
Record Dates: First submitted 2022-03-05; First posted 2022-03-25 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Healthy Aging
Keywords: Dual-Task; Cognitive-Motor Interference; Functional Mobility; Cognition; Motor Performance

STUDY DESIGN:
Intervention Model Description: Subjects are block randomized into 3 parallel groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual Task One (Experimental): Participants perform a cognitive-motor dual-task where the motor task is the same for all groups and the simultaneously performed cognitive task is simple.
  Interventions: Other: Cognitive-motor dual-task
- Dual Task Two (Experimental): Participants perform a cognitive-motor dual-task where the motor task is the same for all groups and the simultaneously performed cognitive task is complex.
  Interventions: Other: Cognitive-motor dual-task
- Control (Active Comparator): Participants perform only a motor-task that is the same for all groups (no simultaneous cognitive task).
  Interventions: Other: Motor Task

INTERVENTIONS:
Other: Motor Task — A visuomotor task is presented where an individual must match their knee to an ellipse that moves up and down on a screen, resulting in a marching-in-place motion at a specified frequency.
  Arms: Control
Other: Cognitive-motor dual-task — While performing the "Motor Task" intervention, letters of different colors and orientation randomly appear one at a time on the screen. During the Cognitive-motor dual-task, individuals are instructed to count the number of times that either 1 (simple cognitive task), or 2 (complex cognitive task) characters appear on the screen during the motor task.
  Arms: Dual Task One; Dual Task Two

SUMMARY:
This study seeks to understand what factors influence the capacity to perform simultaneous motor and cognitive tasks in older adults to improve movement throughout their community with the least risk of injury. To function in the real world, one needs to "walk and talk", or to move about the community while attending to their environment. Navigating a busy environment becomes increasingly difficult due to the multitude of constraints placed on the organism by both the brain and the body that are associated with aging. Resulting lack of movement causes a downward spiral; further decreasing function and increasing risk of co-morbidities. This will impose an enormous cost on our healthcare system as the elderly population continues to grow in the United States. The investigators aim to investigate both cognitive and movement changes during aging to prevent declines in functional mobility. The investigators will do this through eight weeks training of simultaneous cognitive and motor tasks (cognitive-motor training).

DETAILED DESCRIPTION:
In order to functionally move through one's community, it is vital to be able to perform simultaneous motor and cognitive tasks (cognitive-motor dual-task). This allows us to talk to another person, scan the environment for oncoming traffic, and avoid objects that are in our path when walking. This even allows high level sporting participation, such as predicting an opponents' path when sprinting and cutting to score a goal. Unfortunately, aging is associated with increased difficulty in performing cognitive-motor tasks. A classical example is when older adults stop walking in order to talk to another person. Several studies have established that an increase in age is associated with increased cognitive resources required to perform normally automatic motor tasks. Deficits in cognitive-motor dual-task capabilities have been observed not only in older adults, but also in those with neuromuscular compromise due to factors such as stroke and Parkinson's, and even with altered cognition in mild cognitive impairment and Attention Deficit Disorder.

Although these early investigations suggest a relationship between physical and cognitive capabilities, little is known regarding the appropriate level of cognitive task difficulty that will result in improvements or delays in learning a motor task. Conflicting results are noted in the few studies that have investigated this line of research. Some support that a concurrent cognitive task provides a context that facilitates motor learning, while other show that cognitive load prevents individuals from fully learning the motor task . Further, there are very few studies that investigate the effect of cognitive load on the transfer of motor learning to new task conditions for weight-bearing activities. Early evidence suggests that generalizability of learning diminishes the further participants are from the initial task conditions. Interestingly, cognition has been suggested to play a vital role in motor learning, performance, and dual-task capability. Working memory capacity, or the process that allows the maintenance and manipulation of information over a short period of time, has been shown to strongly relate to the rate at which younger adults learn motor sequences, and moderately relate the motor learning of older adults. Executive function, or the properties of cognitive flexibility, problem-solving, and response maintenance, also plays a role in motor learning and performance. Decrements in executive function has been shown to precede mobility limitations, and might even predict gains in mobility from a physical intervention. Executive function may also predict a large portion of the variability when under the context of simultaneously having a cognitive load. There continues to be a lack of understanding of what cognitive capacity is required to perform simultaneous mobility and cognitive tasks with the least risk of injury, and what dose of intervention in both physical and cognitive realms are necessary to induce an improvement in function of both systems.

Purpose: To determine the impact an intervention using simultaneous cognitive and motor tasks on the capacity of healthy adults to improve in functional mobility and cognition.

Research Question: Does a cognitive-motor intervention impact functional mobility and cognition of healthy older adults?

Following obtaining consent from the subject, testing will take place three times a week for 8 weeks. Subjects are randomly assigned to one of each of the three groups: control group, simple cognitive group, or complex cognitive group.

Subjects will be informed that they are randomly assigned to one of three possible groups. Subjects will then be asked to perform either a visuomotor task only (control group), or a visuomotor task with a simultaneous cognitive task (simple cognitive group and complex cognitive group). The visuomotor task is the same regardless of group assignment. The difference in intervention between groups is based on the simultaneous task that the individual will perform: the control group will perform no cognitive task, the simple cognitive group will perform a task of counting a defined letter that appears on the screen, and the complex cognitive group will be assigned the task of counting two assigned letters that appear on the screen. The visuomotor task consists of performing a standing in-place march, lifting alternating knees to 60 degrees of hip flexion, eight cycles on each leg. A custom computer program displays a real-time video of the individual on the screen with an overlay of markers indicating computerized detection (Microsoft Kinect) of the knee joint. A prescribed marching rate is determined by an ellipse on the screen that prescribes the displacement (degrees of hip flexion) and rate of movement (speed) in which to move. Subjects will be allowed light touch for balance if required. One minute of seated rest will be provided between trials with the option of longer rest as needed. Video of the subject is saved in a de-identified format consisting of the view of the individual on the screen and the target task only during the duration of each individual trial. The cognitive task is displayed on the same screen as the motor task. Letters of different orientations and colors appear and disappear on the screen. Each of the 24 sessions will involve performing approximately 20 trials of the visuomotor and cognitive task (control group: visuomotor task only, intervention groups: visuomotor + cognitive task).

Additional details regarding the visuomotor and cognitive tasks are as follows. On the first day, 13th, and 24th days, subjects will perform 20 training trials at a medium speed of the marching task (training), followed by 5 trials of varying marching speeds (testing) by altering the speed (not the amplitude) of a target ellipse that moves on the screen. Then, subjects will be asked to perform one trial of each the simple and the complex cognitive tasks without performing the marching task (cognitive task only). On days 13, and 24 days, subjects will also perform the 5 testing trials under each of the other groups' cognitive task assignment (e.g. a subject assigned to the simple cognitive task group would first perform 5 training and 5 testing trials while performing the simple cognitive task, they would then perform 5 testing trials with the complex cognitive task followed by 5 trials while only performing the motor task). During all other days of the 24 interventions, subjects will perform 20 trials of the medium speed visuomotor task, performing only the cognitive task required of their assigned group.

Additionally, on the 1st,13th, and 24th day, the investigators will take height, weight, and use a scale that measures the participant's body fat percentage (by standing barefoot on the scale). Subjects will be asked to fill out questionnaires which will include information about medical, physical and social life, cognition, activity level, sleep quality and pain levels (see attached forms). Subjects will then be asked to undergo computerized testing of general cognitive function and perceived health via the NIH Toolbox Cognition Battery and PROMIS (via iPad app), and a paper-based assessment of cognition (Montreal Cognitive Assessment). During the NIH Toolbox Cognition Battery test, subjects will sit comfortably in a chair with their arm resting on a table and will perform four tests: the Flanker Inhibitory Control and Attention Test (FLCAT), The List Sorting Working memory Test (LSWMT), The Dimensional Change Card Sort Test (DCCST), and the Processing Speed Test (PST). The FLCAT, DCCST, and PST tests require the user to select an object on the screen using their finger as quickly as possible; the LSWMT will require no movement, but to recite objects of animals and fruits that appear on the screen of the iPad. The Subjects are free to skip any questions or tests that they would prefer not to answer or complete. A test of balance is performed asking the individual to stand on a pressure sensitive mat (Zeno Mat) to record foot pressures and amount of body sway. They will be asked to stand in place with their 1) eyes open, 2) eyes closed, and 3) performing a cognitive task while standing on each foot (single limb stance). Subjects will then be asked to perform a Timed Up and Go (TUG) test under conditions of performing a cognitive task (TUG Cognitive), and without a secondary task (TUG). The TUG test consists of moving as quickly as possible through standing from sitting, walking 3 meters, turning around, and returning three meters to return to the starting seated position. Each test is usually performed in under 30 seconds. Subjects will then be asked to perform a 10-meter walk test, where in the middle of the 8 meters of self-selected walking, they will walk over a pressure sensitive mat (ZenoMat) to determine properties of gait. The 10m walk test will be perform with and without a simultaneous cognitive task at a speed that they feel is normal for them, and then as quickly as they can walk safely.

On days 1, 2, 13, and 24, the investigators will use wireless electrodes with a disposable adhesive interface will be placed over the alcohol abraded skin of lower extremity muscles in order to collect surface electromyography. Following placement of electrodes subjects will be asked to perform three maximal volitional isometric contraction (MVIC) for each muscle. Each MVIC is achieved by the experimenter applying manual resistance in serial with a hand-held dynamometer at the distal most portion of the segment (leg) to which the muscle attaches. The subject is then provided with verbal encouragement to move the limb being tested in the primary direction of muscle movement (eg. For the quadriceps muscles, resistance is applied to the distal tibia at the level of just proximal to the malleoli during knee extension). Between each maximal effort, 1-min rest will be provided to prevent fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Between 60 and 95 Years Old
* Self-described as generally healthy
* Normal or corrected to normal vision
* Able to stand on one foot for at least 3 seconds with minimal sway and no loss of balance

Exclusion Criteria:

* Known neurologic disorder affecting mobility or cognition
* Self-reported known moderate or greater lower extremity arthritis
* Known disease process that affects muscle function
* Color Blindness
* Lower extremity pain in the previous 15 days
* Known learning or attention deficit
* Currently taking medication that affects attention, learning, and/or memory
* Known Cardiovascular Disease of previous heart attack or cardiomyopathy
* Chronic Kidney Disease
* Severe Obesity as defined by a BMI of greater than or equal to 40 Kg/m2

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Change in Timed Up and Go Tests in 4 week increments | Baseline, Week 4, and Week 8
  Timed Up and Go, and Timed Up and Go Cognitive
Change in 10 meter walk test self-selected pace in 4 week increments | Baseline, Week 4, and Week 8
  self selected pace walking over an instrumented mat (ZenoMat) both single task and while counting serial 3's
Change in Cognition in 4 week increments | Baseline, Week 4, and Week 8
  Components of Cognitive Fluidity as measured by the NIH Toolbox Cognitive Battery

SECONDARY OUTCOMES:
Balance Test Performance in 4 week increments | Baseline, Week 4, and Week 8
  Single Leg Stand with and without Cognitive Task
change in 10 meter walk test fast pace in 4 week increments | Baseline, Week 4, and Week 8
  Walking as fast as possible without running an instrumented mat (ZenoMat) both single task and while counting serial 3's
Change in Muscle Electromyography in 4 week increments | Baseline, Week 4 and Week 8
  Surface electromyography (sEMG) will be obtained by placing wireless Delsys Trigno electrodes on the skin over the muscles of the lower extremities (tibialis anterior, lateral gastrocnemius, Rectus Femoris, Vastus Medialis, Lateral Hamstrings, and Gluteus Maximus). EMG will used to measure muscle activity during the cognitive-motor dual-task in order to measure changes in neuromuscular control strategy as subjects learn to perform the task.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Cole, DPT, Ph. D., Principal Investigator — The George Washington University
Locations (1):
- The George Washington University, Department of Health, Human Function and Rehabilitation Science, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] Alcock L, Galna B, Lord S, Rochester L. Characterisation of foot clearance during gait in people with early Parkinson׳s disease: Deficits associated with a dual task. J Biomech. 2016 Sep 6;49(13):2763-2769. doi: 10.1016/j.jbiomech.2016.06.007. Epub 2016 Jun 15. PMID 27363617
- [Background] Alvarez JA, Emory E. Executive function and the frontal lobes: a meta-analytic review. Neuropsychol Rev. 2006 Mar;16(1):17-42. doi: 10.1007/s11065-006-9002-x. PMID 16794878
- [Background] Alves FD, Souza GC, Biolo A, Clausell N. Comparison of two bioelectrical impedance devices and dual-energy X-ray absorptiometry to evaluate body composition in heart failure. J Hum Nutr Diet. 2014 Dec;27(6):632-8. doi: 10.1111/jhn.12218. Epub 2014 Mar 29. PMID 24684316
- [Background] Amboni M, Barone P, Iuppariello L, Lista I, Tranfaglia R, Fasano A, Picillo M, Vitale C, Santangelo G, Agosti V, Iavarone A, Sorrentino G. Gait patterns in Parkinsonian patients with or without mild cognitive impairment. Mov Disord. 2012 Oct;27(12):1536-43. doi: 10.1002/mds.25165. Epub 2012 Oct 2. PMID 23032876
- [Background] Baddeley A, Logie R, Bressi S, Della Sala S, Spinnler H. Dementia and working memory. Q J Exp Psychol A. 1986 Nov;38(4):603-18. doi: 10.1080/14640748608401616. No abstract available. PMID 3809575
- [Background] Baetens T, De Kegel A, Palmans T, Oostra K, Vanderstraeten G, Cambier D. Gait analysis with cognitive-motor dual tasks to distinguish fallers from nonfallers among rehabilitating stroke patients. Arch Phys Med Rehabil. 2013 Apr;94(4):680-6. doi: 10.1016/j.apmr.2012.11.023. Epub 2012 Nov 24. PMID 23187040
- [Background] Balady GJ, Arena R, Sietsema K, Myers J, Coke L, Fletcher GF, Forman D, Franklin B, Guazzi M, Gulati M, Keteyian SJ, Lavie CJ, Macko R, Mancini D, Milani RV; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Interdisciplinary Council on Quality of Care and Outcomes Research. Clinician's Guide to cardiopulmonary exercise testing in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 13;122(2):191-225. doi: 10.1161/CIR.0b013e3181e52e69. Epub 2010 Jun 28. No abstract available. PMID 20585013
- [Background] Beaver WL, Wasserman K, Whipp BJ. A new method for detecting anaerobic threshold by gas exchange. J Appl Physiol (1985). 1986 Jun;60(6):2020-7. doi: 10.1152/jappl.1986.60.6.2020. PMID 3087938
- [Background] Bedard P, Song JH. Attention modulates generalization of visuomotor adaptation. J Vis. 2013 Oct 16;13(12):12. doi: 10.1167/13.12.12. PMID 24133292
- [Background] Blumen HM, Holtzer R, Brown LL, Gazes Y, Verghese J. Behavioral and neural correlates of imagined walking and walking-while-talking in the elderly. Hum Brain Mapp. 2014 Aug;35(8):4090-104. doi: 10.1002/hbm.22461. Epub 2014 Feb 12. PMID 24522972
- [Background] Bo J, Borza V, Seidler RD. Age-related declines in visuospatial working memory correlate with deficits in explicit motor sequence learning. J Neurophysiol. 2009 Nov;102(5):2744-54. doi: 10.1152/jn.00393.2009. Epub 2009 Sep 2. PMID 19726728
- [Background] Bo J, Seidler RD. Visuospatial working memory capacity predicts the organization of acquired explicit motor sequences. J Neurophysiol. 2009 Jun;101(6):3116-25. doi: 10.1152/jn.00006.2009. Epub 2009 Apr 8. PMID 19357338
- [Background] Bolanowski M, Nilsson BE. Assessment of human body composition using dual-energy x-ray absorptiometry and bioelectrical impedance analysis. Med Sci Monit. 2001 Sep-Oct;7(5):1029-33. PMID 11535954
- [Background] Brauer SG, Morris ME. Can people with Parkinson's disease improve dual tasking when walking? Gait Posture. 2010 Feb;31(2):229-33. doi: 10.1016/j.gaitpost.2009.10.011. Epub 2009 Dec 6. PMID 19969461
- [Background] Cockburn J, Haggard P, Cock J, Fordham C. Changing patterns of cognitive-motor interference (CMI) over time during recovery from stroke. Clin Rehabil. 2003 Mar;17(2):167-73. doi: 10.1191/0269215503cr597oa. PMID 12625657
- [Background] Dennis A, Dawes H, Elsworth C, Collett J, Howells K, Wade DT, Izadi H, Cockburn J. Fast walking under cognitive-motor interference conditions in chronic stroke. Brain Res. 2009 Sep 1;1287:104-10. doi: 10.1016/j.brainres.2009.06.023. Epub 2009 Jun 13. PMID 19527695
- [Background] Doi T, Makizako H, Shimada H, Park H, Tsutsumimoto K, Uemura K, Suzuki T. Brain activation during dual-task walking and executive function among older adults with mild cognitive impairment: a fNIRS study. Aging Clin Exp Res. 2013 Oct;25(5):539-44. doi: 10.1007/s40520-013-0119-5. Epub 2013 Aug 15. PMID 23949972
- [Background] Elovainio M, Kivimaki M, Ferrie JE, Gimeno D, De Vogli R, Virtanen M, Vahtera J, Brunner EJ, Marmot MG, Singh-Manoux A. Physical and cognitive function in midlife: reciprocal effects? A 5-year follow-up of the Whitehall II study. J Epidemiol Community Health. 2009 Jun;63(6):468-73. doi: 10.1136/jech.2008.081505. PMID 19439578
- [Background] Erickson KI, Colcombe SJ, Wadhwa R, Bherer L, Peterson MS, Scalf PE, Kramer AF. Neural correlates of dual-task performance after minimizing task-preparation. Neuroimage. 2005 Dec;28(4):967-79. doi: 10.1016/j.neuroimage.2005.06.047. Epub 2005 Aug 16. PMID 16109493
- [Background] Fritz NE, Cheek FM, Nichols-Larsen DS. Motor-Cognitive Dual-Task Training in Persons With Neurologic Disorders: A Systematic Review. J Neurol Phys Ther. 2015 Jul;39(3):142-53. doi: 10.1097/NPT.0000000000000090. PMID 26079569
- [Background] Galna B, Lord S, Rochester L. Is gait variability reliable in older adults and Parkinson's disease? Towards an optimal testing protocol. Gait Posture. 2013 Apr;37(4):580-5. doi: 10.1016/j.gaitpost.2012.09.025. Epub 2012 Oct 25. PMID 23103242
- [Background] Goh HT, Sullivan KJ, Gordon J, Wulf G, Winstein CJ. Dual-task practice enhances motor learning: a preliminary investigation. Exp Brain Res. 2012 Oct;222(3):201-10. doi: 10.1007/s00221-012-3206-5. Epub 2012 Aug 12. PMID 22886044
- [Background] Gothe K, Oberauer K, Kliegl R. Age differences in dual-task performance after practice. Psychol Aging. 2007 Sep;22(3):596-606. doi: 10.1037/0882-7974.22.3.596. PMID 17874957
- [Background] Gothe NP, Fanning J, Awick E, Chung D, Wojcicki TR, Olson EA, Mullen SP, Voss M, Erickson KI, Kramer AF, McAuley E. Executive function processes predict mobility outcomes in older adults. J Am Geriatr Soc. 2014 Feb;62(2):285-90. doi: 10.1111/jgs.12654. Epub 2014 Jan 21. PMID 24521364
- [Background] Herath P, Klingberg T, Young J, Amunts K, Roland P. Neural correlates of dual task interference can be dissociated from those of divided attention: an fMRI study. Cereb Cortex. 2001 Sep;11(9):796-805. doi: 10.1093/cercor/11.9.796. PMID 11532885
- [Background] Jacobs JV, Nutt JG, Carlson-Kuhta P, Allen R, Horak FB. Dual tasking during postural stepping responses increases falls but not freezing in people with Parkinson's disease. Parkinsonism Relat Disord. 2014 Jul;20(7):779-81. doi: 10.1016/j.parkreldis.2014.04.001. Epub 2014 Apr 14. PMID 24768615
- [Background] Jones AM, Carter H. The effect of endurance training on parameters of aerobic fitness. Sports Med. 2000 Jun;29(6):373-86. doi: 10.2165/00007256-200029060-00001. PMID 10870864
- [Background] Kafri MW, Potter JF, Myint PK. Multi-frequency bioelectrical impedance analysis for assessing fat mass and fat-free mass in stroke or transient ischaemic attack patients. Eur J Clin Nutr. 2014 Jun;68(6):677-82. doi: 10.1038/ejcn.2013.266. Epub 2014 Jan 8. PMID 24398644
- [Background] Leitner Y, Barak R, Giladi N, Peretz C, Eshel R, Gruendlinger L, Hausdorff JM. Gait in attention deficit hyperactivity disorder : effects of methylphenidate and dual tasking. J Neurol. 2007 Oct;254(10):1330-8. doi: 10.1007/s00415-006-0522-3. Epub 2007 Apr 2. PMID 17401735
- [Background] Lundin-Olsson L, Nyberg L, Gustafson Y. "Stops walking when talking" as a predictor of falls in elderly people. Lancet. 1997 Mar 1;349(9052):617. doi: 10.1016/S0140-6736(97)24009-2. No abstract available. PMID 9057736
- [Background] Makizako H, Doi T, Shimada H, Yoshida D, Takayama Y, Suzuki T. Relationship between dual-task performance and neurocognitive measures in older adults with mild cognitive impairment. Geriatr Gerontol Int. 2013 Apr;13(2):314-21. doi: 10.1111/j.1447-0594.2012.00898.x. Epub 2012 Jun 14. PMID 22694665
- [Background] Makizako H, Doi T, Shimada H, Yoshida D, Tsutsumimoto K, Uemura K, Suzuki T. Does a multicomponent exercise program improve dual-task performance in amnestic mild cognitive impairment? A randomized controlled trial. Aging Clin Exp Res. 2012 Dec;24(6):640-6. doi: 10.3275/8760. Epub 2012 Nov 26. PMID 23211228
- [Background] Marques NR, Hallal CZ, Spinoso DH, Morcelli MH, Crozara LF, Goncalves M. Applying different mathematical variability methods to identify older fallers and non-fallers using gait variability data. Aging Clin Exp Res. 2017 Jun;29(3):473-481. doi: 10.1007/s40520-016-0592-8. Epub 2016 Jun 2. PMID 27256077
- [Background] Muir SW, Speechley M, Wells J, Borrie M, Gopaul K, Montero-Odasso M. Gait assessment in mild cognitive impairment and Alzheimer's disease: the effect of dual-task challenges across the cognitive spectrum. Gait Posture. 2012 Jan;35(1):96-100. doi: 10.1016/j.gaitpost.2011.08.014. Epub 2011 Sep 22. PMID 21940172
- [Background] O'Shea S, Morris ME, Iansek R. Dual task interference during gait in people with Parkinson disease: effects of motor versus cognitive secondary tasks. Phys Ther. 2002 Sep;82(9):888-97. PMID 12201803
- [Background] Plummer P, Eskes G. Measuring treatment effects on dual-task performance: a framework for research and clinical practice. Front Hum Neurosci. 2015 Apr 28;9:225. doi: 10.3389/fnhum.2015.00225. eCollection 2015. PMID 25972801
- [Background] Plummer P, Eskes G, Wallace S, Giuffrida C, Fraas M, Campbell G, Clifton KL, Skidmore ER; American Congress of Rehabilitation Medicine Stroke Networking Group Cognition Task Force. Cognitive-motor interference during functional mobility after stroke: state of the science and implications for future research. Arch Phys Med Rehabil. 2013 Dec;94(12):2565-2574.e6. doi: 10.1016/j.apmr.2013.08.002. Epub 2013 Aug 20. PMID 23973751
- [Background] Plummer P, Iyigun G. Effects of Physical Exercise Interventions on Dual-Task Gait Speed Following Stroke: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2018 Dec;99(12):2548-2560. doi: 10.1016/j.apmr.2018.04.009. Epub 2018 May 5. PMID 29738743
- [Background] Plummer P, Osborne MB. What Are We Attempting to Improve When We Train Dual-Task Performance? J Neurol Phys Ther. 2015 Jul;39(3):154-5. doi: 10.1097/NPT.0000000000000097. No abstract available. PMID 26050072
- [Background] Plummer P, Zukowski LA, Giuliani C, Hall AM, Zurakowski D. Effects of Physical Exercise Interventions on Gait-Related Dual-Task Interference in Older Adults: A Systematic Review and Meta-Analysis. Gerontology. 2015;62(1):94-117. doi: 10.1159/000371577. Epub 2015 Feb 19. PMID 25721432
- [Background] Roche RA, Commins S, Agnew F, Cassidy S, Corapi K, Leibbrand S, Lipson Z, Rickard J, Sorohan J, Wynne C, O'Mara SM. Concurrent task performance enhances low-level visuomotor learning. Percept Psychophys. 2007 May;69(4):513-22. doi: 10.3758/bf03193908. PMID 17727104
- [Background] Sanli EA, Lee TD. What roles do errors serve in motor skill learning? An examination of two theoretical predictions. J Mot Behav. 2014;46(5):329-37. doi: 10.1080/00222895.2014.913544. Epub 2014 May 23. PMID 24857405
- [Background] Shorer Z, Becker B, Jacobi-Polishook T, Oddsson L, Melzer I. Postural control among children with and without attention deficit hyperactivity disorder in single and dual conditions. Eur J Pediatr. 2012 Jul;171(7):1087-94. doi: 10.1007/s00431-012-1695-7. Epub 2012 Feb 16. PMID 22350284
- [Background] Song JH, Bedard P. Paradoxical benefits of dual-task contexts for visuomotor memory. Psychol Sci. 2015 Feb;26(2):148-58. doi: 10.1177/0956797614557868. Epub 2014 Dec 10. PMID 25501806
- [Background] Strobach T, Frensch P, Muller H, Schubert T. Age- and practice-related influences on dual-task costs and compensation mechanisms under optimal conditions of dual-task performance. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2012;19(1-2):222-47. doi: 10.1080/13825585.2011.630973. Epub 2011 Dec 14. PMID 22168474
- [Background] Strobach T, Frensch PA, Soutschek A, Schubert T. Investigation on the improvement and transfer of dual-task coordination skills. Psychol Res. 2012 Nov;76(6):794-811. doi: 10.1007/s00426-011-0381-0. Epub 2011 Sep 27. PMID 21947746
- [Background] Svendsen OL, Haarbo J, Heitmann BL, Gotfredsen A, Christiansen C. Measurement of body fat in elderly subjects by dual-energy x-ray absorptiometry, bioelectrical impedance, and anthropometry. Am J Clin Nutr. 1991 May;53(5):1117-23. doi: 10.1093/ajcn/53.5.1117. PMID 2021122
- [Background] Woollacott M, Shumway-Cook A. Attention and the control of posture and gait: a review of an emerging area of research. Gait Posture. 2002 Aug;16(1):1-14. doi: 10.1016/s0966-6362(01)00156-4. PMID 12127181
- [Background] Wu T, Liu J, Hallett M, Zheng Z, Chan P. Cerebellum and integration of neural networks in dual-task processing. Neuroimage. 2013 Jan 15;65:466-75. doi: 10.1016/j.neuroimage.2012.10.004. Epub 2012 Oct 11. PMID 23063842
- [Background] (2004). Oxygen Uptake Kinetics in Sport, Exercise and Medicine, Routledge.
- [Background] Dalleck, L.C. and J.S. Tischendorf. Guidelines for Exercise Testing and Prescription (ACSM). Encyclopedia of Lifestyle Medicine & Health, SAGE Publications, Inc.
- [Background] Wajda DA, Mirelman A, Hausdorff JM, Sosnoff JJ. Intervention modalities for targeting cognitive-motor interference in individuals with neurodegenerative disease: a systematic review. Expert Rev Neurother. 2017 Mar;17(3):251-261. doi: 10.1080/14737175.2016.1227704. Epub 2016 Sep 12. PMID 27548008
- [Background] Cole KR, Shields RK. Age and Cognitive Stress Influences Motor Skill Acquisition, Consolidation, and Dual-Task Effect in Humans. J Mot Behav. 2019;51(6):622-639. doi: 10.1080/00222895.2018.1547893. Epub 2019 Jan 2. PMID 30600778